CLINICAL TRIAL: NCT02515617
Title: Drainage of Subglottic Secretions and Prevention of Ventilator-associated Pneumonia in Intensive carE Units: Medico-Economic Study With a Randomized clusTer and crossovER Design: DEMETER Study
Brief Title: Medico-economic Study of the Subglottic Secretions Drainage in Prevention of Ventilator-associated Pneumonia (DEMETER)
Acronym: DEMETER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); URC Eco Ile de France (Unknown); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CHD 045-14
Record Dates: First submitted 2015-07-31; First posted 2015-08-05 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2018-01

CONDITIONS: Ventilator-associated Pneumonia
Keywords: Ventilator-associated pneumonia; Subglottic-secretions drainage; Critically ill patients; Cost-utility analysis; Prevention
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period with endotracheal tubes not allowing SSD (Active Comparator): During this period, patients will be intubated with standard endotracheal tubes not allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes not allowing SSD
- Period with endotracheal tubes allowing SSD (Experimental): During this period, patients will be intubated with specific endotracheal tubes allowing Subglottic Secretions Drainage
  Interventions: Device: Endotracheal tubes allowing SSD

INTERVENTIONS:
Device: Endotracheal tubes not allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure
  Arms: Period with endotracheal tubes not allowing SSD
Device: Endotracheal tubes allowing SSD — In each participating center, a bundle of VAP prevention will be applied: elevate the head of the bed to 30°-45°, regular oral care, manage patients with sedation algorithm, assess readiness to extubate daily, intermittent control of endotracheal tube cuff pressure.
  In addition, SSD will be realized using a 10 ml syringe at in attending frequency of 2 hours.
  Arms: Period with endotracheal tubes allowing SSD

SUMMARY:
In France, despite the implementation of bundles to prevent Ventilator-Associated Pneumonia (VAP) in the last decades, the VAP incidence remains high above 10 per cent. In the last american recommendations of VAP prevention, the drainage of subglottic secretions (SSD) has been notified among the "basic practices" to prevent VAP. Nevertheless, the diffusion of SSD in ICUs remains limited. This situation is largely due to the initial overcost of the specific endotracheal tubes allowing SSD and to the unavailability of these devices in medical units in which patients are intubated before the ICU admission. So, this pragmatical cluster randomized and cross-over study evaluates the medico-economic impact of the subglottic secretions drainage in addition to VAP prevention bundles in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Invasive mechanical ventilation delivered via an endotracheal tube and expected to be required more than 24 hours
* Intubation performed in units in which the specific endotracheal tube allowing the subglottic secretions drainage (SSD) will be available during the SSD period of the trial
* Information delivered

Exclusion Criteria:

* Previous inclusion in the study
* Patients moribund at the ICU admission
* Pregnant, parturient or breast-feeding woman
* Patient hospitalized without consent and/or deprived of liberty by court's decision
* Patient under guardianship or curators
* Lack of social insurance
* Concomitant inclusion in a trial on VAP prevention
* Patient with no comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2577 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Incremental cost-utility ratio | 1 year after ICU admission
  Incremental cost to gain an extra quality-adjusted life-year (QALY) with the SSD implementation

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio | 1 year after ICU admission
  Incremental cost to gain an additional patient free of adjudicated VAP
Incremental cost-utility ratio (subgroup analysis) | 1 year after ICU admission
  Incremental cost to gain an extra quality-adjusted life-year (QALY) with the SSD in considering patients alive at the ICU discharge
Incremental cost-effectiveness ratio | 1 year after ICU admission
  Incremental cost to gain an additional life-year
Budget impact analysis | 5 years
Microbiologically-confirmed VAP incidence | 90 days after the start of invasive mechanical ventilation
Microbiologically-confirmed VAP density of incidence | 90 days after the start of invasive mechanical ventilation
Defined Daily Dose of antibiotics consumption | Until discharge from ICU, an expected average of 12 days
Ventilator-associated Conditions incidence | 90 days after the start of invasive mechanical ventilation
Ventilator-associated Conditions density of incidence | 90 days after the start of invasive mechanical ventilation
Infection related Ventilator-associated Conditions incidence | 90 days after the start of invasive mechanical ventilation
Duration of invasive mechanical ventilation | Until weaning of mechanical ventilation, an expected average of 10 days
Ventilator-free days | 90 days after the start of invasive mechanical ventilation
ICU length of stay | Until discharge from ICU, an expected average of 12 days
Hospital length of stay | Until discharge from hospital, an expected average of 20 days
ICU mortality | Until discharge from ICU, an expected average of 12 days
90-days mortality | 90 days after ICU admission
180-days mortality | 180 days after ICU admission
1 year mortality | 1 year after ICU admission
Post-extubation laryngo-tracheal dyspnea incidence | Until weaning of mechanical ventilation,, an expected average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude LACHERADE, MD, Principal Investigator — CHD VENDEE
Locations (25):
- CHU André Vésale ,, Montigny-le-Tilleul, Belgium
- France (21):
  - CH Angoulème, Angoulème
  - CH Annecy Genevois, Annecy
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Intercommunal des Portes de l'Oise, Beaumont-sur-Oise
  - CHU Dijon, Dijon
  - CHD Vendee, La Roche-sur-Yon
  - CH Docteur Schaffner, Lens
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - CHU marseilles, Hôpital Nord, Marseilels
  - CH de Montauban, Montauban
  - CHU Nantes, Nantes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - CHI Poissy Saint Germain, Poissy
  - CHU Poitiers, Poitiers
  - Centre Hospitalier René Dubos, Pontoise
  - Hôpital Delafontaine, Saint-Denis
  - CH de Saint Nazaire, Saint-Nazaire
  - CHU de Strasbourg Hôpital de Hautepierre, Strasbourg
  - CHU de Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CHU Tours, site Bretonneau, Tours
  - CHU Tours, site Trousseau, Tours
- CHU Pointe à Pitre les Abymes, Pointe-à-Pitre, Guadeloupe
- Reunion (2):
  - CHU La Réunion, site de Saint Denis de la Réunion, Saint-Denis
  - CHU La Réunion, site de Saint Pierre de la Réunion, Saint-Pierre

REFERENCES:
- [Background] Muscedere J, Rewa O, McKechnie K, Jiang X, Laporta D, Heyland DK. Subglottic secretion drainage for the prevention of ventilator-associated pneumonia: a systematic review and meta-analysis. Crit Care Med. 2011 Aug;39(8):1985-91. doi: 10.1097/CCM.0b013e318218a4d9. PMID 21478738
- [Background] Lacherade JC, De Jonghe B, Guezennec P, Debbat K, Hayon J, Monsel A, Fangio P, Appere de Vecchi C, Ramaut C, Outin H, Bastuji-Garin S. Intermittent subglottic secretion drainage and ventilator-associated pneumonia: a multicenter trial. Am J Respir Crit Care Med. 2010 Oct 1;182(7):910-7. doi: 10.1164/rccm.200906-0838OC. Epub 2010 Jun 3. PMID 20522796
- [Background] Klompas M, Branson R, Eichenwald EC, Greene LR, Howell MD, Lee G, Magill SS, Maragakis LL, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia in acute care hospitals: 2014 update. Infect Control Hosp Epidemiol. 2014 Sep;35 Suppl 2:S133-54. doi: 10.1017/s0899823x00193894. No abstract available. PMID 25376073
- [Background] Branch-Elliman W, Wright SB, Howell MD. Determining the Ideal Strategy for Ventilator-associated Pneumonia Prevention. Cost-Benefit Analysis. Am J Respir Crit Care Med. 2015 Jul 1;192(1):57-63. doi: 10.1164/rccm.201412-2316OC. PMID 25871807
- [Background] Loupec T, Petitpas F, Kalfon P, Mimoz O. Subglottic secretion drainage in prevention of ventilator-associated pneumonia: mind the gap between studies and reality. Crit Care. 2013 Dec 9;17(6):R286. doi: 10.1186/cc13149. No abstract available. PMID 24321315